CLINICAL TRIAL: NCT04325984
Title: Ruolo Del Desametasone Per il Controllo Multimodale Del Dolore Postoperatorio in Chirurgia Toracica
Brief Title: Role of Dexamethasone in Multimodal Analgesia for Postoperative Pain in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Marzia Umari, Principal Investigator, University of Trieste
Other Study IDs: 173_2018_DexaPOP
Record Dates: First submitted 2020-03-14; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Dexamethasone Adverse Reaction; Postoperative Pain; Postoperative Thoracic Procedure Complication; Analgesia
Keywords: Thoracic surgery; Postoperative complications; Dexamethasone; Postoperative Nausea and Vomiting; Hyperglycaemia; Video Assisted ThoracoScopy (VATS); Multimodal Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Postoperative Complications; Postoperative Nausea and Vomiting; Hyperglycemia | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dexamethasone group: Group of patients receiving dexamethasone 8 mg as part of the multimodal analgesia.
  Interventions: Drug: Dexamethasone
- Control group: Group of patients receiving multimodal analgesia, not comprising dexamethasone; moreover, ondansetron 4 mg is administered for the control of PONV.

INTERVENTIONS:
Drug: Dexamethasone — To the Dexamethasone group, at the moment of the induction of anaesthesia, dexamethasone 8 mg is administered.
  Groups: Dexamethasone group

SUMMARY:
The aim of the study is to evaluate the analgesic properties of dexamethasone and to quantify the possible associated postoperative complications, such as wound infections and hyperglycaemia, in patients who underwent lobectomy, segmentectomy or atypical resection surgery with a mini-thoracotomy approach or video-assisted thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
We designed an observational study, aimed to evaluate the possible reduction in morphine consumption in thoracic patients, who were administered dexamethasone compared to who didn't received the drug.

The research wants to assess the presence of additional analgesic properties, besides the well known antiemetic effect, in the intraoperative administration of dexamethasone, and the possible postoperative complications, such as wound infections and hyperglycaemia.

The rational is to ameliorate the anaesthesiological management, in particular with a view to a opioid-sparing analgesia in thoracic patients.

To do so, we enrolled thoracic patients, who underwent elective lobectomy, segmentectomy or atypical resection surgery with a mini-thoracotomy approach or video-assisted thoracoscopic surgery (VATS).

We selected two groups: one in which patients were administered dexamethasone 8 mg at the moment of induction, and the other one in which patients didn't received dexamethasone, but ondansetron 4 mg at the end of surgery. Both groups received other antiemetic drugs based on Apfel score and multimodal analgesia, comprising loco-regional analgesia, opioids and other analgesic drugs administration.

The we checked morphine consumption and Numerical Rating Scale (NRS) values for pain in the first 24 hours after surgery.

Moreover we evaluate Post-Operative Nausea and Vomiting (PONV), intra- and post-operative blood glucose levels and wound infection.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m2
* ASA I-III
* Lobectomy, segmentectomy or atypical resection surgery with a mini-thoracotomy approach or VATS

Exclusion Criteria:

* Refusal by the patient to participate or patient unable to express his own consent
* Chronic therapy with medium-high doses of corticosteroids
* Chronic therapy with opioids
* METS ≤ 4, defining an overall decreased cardiovascular fitness
* Urgent or emergency surgery
* Allergy to the active ingredient of the drug used
* Kidney failure at stage III or more
* Liver failure
* Pregnancy
* Drug addiction, patients with a history of drug abuse
* Corrected Qt interval (QTc) > 0,45 for males and 0,47 for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted at our surgical center who underwent elective lobectomy, segmentectomy or atypical resection surgery with a mini-thoracotomy approach or VATS.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours after surgery
  Morphine dose, in milligrams, administered in the 24 hours after the surgery

SECONDARY OUTCOMES:
Static and dynamic Numeric Rating Scale (NRS) | 24 hours after surgery
  Evaluation of Numeric Rating Scale (NRS) for static and dynamic pain; the NRS uses scores from 0 (no pain) to 10 (worst possible pain)

OTHER OUTCOMES:
Glycemic changes | 24 hours after surgery
  Evaluation of intraoperative and postoperative blood glucose levels
Surgical wound infection | At hospital discharge/ at first medical check if discharge was earlier than 7 days
  Evaluation of infectious complication after surgery: assessment of the presence of signs and symptoms of infection of the surgical wound
Postoperative Nausea and Vomiting (PONV) | 24 hours after surgery
  Evaluation of development of postoperative nausea or vomiting, reporting the presence of episodes of nausea or vomiting in the 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Lucangelo, MD PhD, Study Director — University of Trieste; Marzia Umari, MD, Principal Investigator — University of Trieste
Locations (1):
- Cattinara Hospital, Trieste, Italy

REFERENCES:
- [Background] Wenk M, Schug SA. Perioperative pain management after thoracotomy. Curr Opin Anaesthesiol. 2011 Feb;24(1):8-12. doi: 10.1097/ACO.0b013e3283414175. PMID 21084984
- [Background] Doan LV, Augustus J, Androphy R, Schechter D, Gharibo C. Mitigating the impact of acute and chronic post-thoracotomy pain. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):1048-56. doi: 10.1053/j.jvca.2014.02.021. No abstract available. PMID 25107721
- [Background] Henzi I, Walder B, Tramer MR. Dexamethasone for the prevention of postoperative nausea and vomiting: a quantitative systematic review. Anesth Analg. 2000 Jan;90(1):186-94. doi: 10.1097/00000539-200001000-00038. PMID 10625002
- [Background] Waldron NH, Jones CA, Gan TJ, Allen TK, Habib AS. Impact of perioperative dexamethasone on postoperative analgesia and side-effects: systematic review and meta-analysis. Br J Anaesth. 2013 Feb;110(2):191-200. doi: 10.1093/bja/aes431. Epub 2012 Dec 5. PMID 23220857
- [Background] Kakodkar PS. Routine use of dexamethasone for postoperative nausea and vomiting: the case for. Anaesthesia. 2013 Sep;68(9):889-91. doi: 10.1111/anae.12308. Epub 2013 Jul 15. No abstract available. PMID 23848292
- [Background] Standards of Medical Care in Diabetes-2016: Summary of Revisions. Diabetes Care. 2016 Jan;39 Suppl 1:S4-5. doi: 10.2337/dc16-S003. No abstract available. PMID 26696680
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Wenk+M%2C+Schug+SA.+Perioperative+pain+management+after+thoracotomy.+Curr+Opin+Anaesthesiol.+2011+Feb%3B24(1)%3A8%E2%80%9312.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Doan+LV%2C+Augustus+J%2C+Androphy+R%2C+Schechter+D%2C+Gharibo+C.+Mitigating+the+impact+of+acute+and+chronic+post-thoracotomy+pain.+J+Cardiothorac+Vasc+Anesth.+2014+Aug%3B28(4)%3A1048%E2%80%9356.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Henzi+I%2C+Walder+B%2C+Tram%C3%A8r+MR.+Dexamethasone+for+the+prevention+of+postoperative+nausea+and+vomiting%3A+a+quantitative+systematic+review.+Anesth+Analg.+2000+Jan%3B90(1)%3A186%E2%80%9394.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Waldron+NH%2C+Jones+CA%2C+Gan+TJ%2C+Allen+TK%2C+Habib+AS.+Impact+of+perioperative+dexamethasone+on+postoperative+analgesia+and+side-effects%3A+systematic+review+and+meta-analysis.+Br+J+Anaesth.+2012%3B110(2)%3A191%E2%80%93200.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Kakodkar+PS.+Routine+use+of+dexamethasone+for+postoperative+nausea+and+vomiting%3A+the+case+for.+Anaesthesia.+2013+Sep%3B68(9)%3A889%E2%80%9391.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Standards+of+Medical+Care+in+Diabetes%E2%80%942016%3A+Summary+of+Revisions.+Diabetes+Care.+2016+Jan+1%3B39